CLINICAL TRIAL: NCT05213494
Title: A Randomized, Controlled, Crossover Study to Assess the Effects of Soluble Corn Fiber on Gastrointestinal Tolerance and Fecal Microbiome in Healthy Children
Brief Title: The Effects of Soluble Corn Fiber on Gastrointestinal Tolerance and Fecal Microbiome in Healthy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tate & Lyle (Industry)
Collaborators: Biofortis Innovation Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: BIO-2108
Record Dates: First submitted 2021-12-30; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Gastrointestinal Tolerance
Keywords: digestion, fiber, tolerance,
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Low-dose inulin (Active Comparator): 3-5 years old: 3g of fiber/day from inulin mixed in a beverage 6-9 years old: 5g of fiber/day from inulin mixed in a beverage
  Interventions: Other: Inulin
- Low-dose soluble corn fiber (Experimental): 3-5 years old: 3g of fiber/day from soluble corn fiber mixed in a beverage 6-9 years old: 5g of fiber/day from soluble corn fiber mixed in a beverage
  Interventions: Other: soluble corn fiber
- High-dose inulin (Active Comparator): 3-5 years old: 6g of fiber/day from inulin mixed in a beverage 6-9 years old: 8g of fiber/day from inulin mixed in a beverage
  Interventions: Other: Inulin
- High-dose soluble corn fiber (Experimental): 3-5 years old: 6g of fiber/day from soluble corn fiber mixed in a beverage 6-9 years old: 8g of fiber/day from soluble corn fiber mixed in a beverage
  Interventions: Other: soluble corn fiber
- Baseline (No Intervention): 3-9 years old: pre-intervention.

INTERVENTIONS:
Other: Inulin — Inulin, a dietary fiber, will be given in a beverage daily in doses 3g, 5g, 6g, or 8g dependent on arm and age of participants.
  Arms: High-dose inulin; Low-dose inulin
Other: soluble corn fiber — soluble corn fiber, a dietary fiber, will be given in a beverage daily in doses 3g, 5g, 6g, or 8g dependent on arm and age of participants.
  Arms: High-dose soluble corn fiber; Low-dose soluble corn fiber

SUMMARY:
The purpose of this study is to compare the effects of PROMITOR® Soluble Corn Fiber versus inulin on GI symptoms (tolerance), stool consistency (laxation) and fecal microbiome at levels that could contribute to closing the fiber gap. The dose response effects of PROMITOR® Soluble Corn Fiber in healthy children will also be compared.

DETAILED DESCRIPTION:
After initial site visits and randomization children were given a packet of powdered fiber to be mixed into a beverage daily. There were four test arms, described elsewhere. Each study arm lasted 10 days with an 18 day washout in between study periods.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 3-9 years of age, inclusive at Visit 1 (Day -7)
2. Potty trained
3. Bowel movement at least every other day.
4. Regularly consumes breakfast (at least 5 times/week) and agrees to consume breakfast every day during each test period.
5. Willing to maintain physical activity and exercise patterns, body weight, and habitual diet throughout the trial.
6. Willing to refrain from exclusionary medications, supplements, and products throughout the study.
7. No health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history.
8. Caregiver understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator and subject provides informed assent.

Exclusion criteria

1. Regular (>2/week) moderate to severe GI symptoms (as reported by subject and/or caregiver at Visit 1, Day -7). Mild and infrequent (≤ 2/week) GI symptoms are allowed.
2. Subject will be away from caregiver for more than 1 day during the 3-day baseline period (Days -3, -2, and -1) and >48 consecutive hours during the 10 days of study product consumption during each test period. Goal is to recruit subjects who will be with their caregiver all or most of the time to minimize missing data.
3. Clinically important GI conditions that would potentially interfere with the evaluation of the study product [e.g., inflammatory bowel disease, irritable bowel syndrome, gastric reflux, indigestion, dyspepsia, Crohn's disease, celiac disease, gastroparesis, and clinically significant lactose and gluten intolerance or other food or ingredient allergies which includes allergies to milk, eggs, peanuts, tree nuts, wheat and soy (Appendix 9)].
4. Recent (within 2 weeks of Visit 1; Day -7) history of an episode of acute GI illness such as nausea/vomiting or diarrhea (defined as ≥ 3 loose or liquid stools/day).
5. Caregiver-reported history (within 4 weeks of Visit 1; Day -7) of any constipation (<3 bowel movement/week) and diarrhea (≥3 of more loose stools/day) at the discretion of the Clinical Investigator.
6. Uncontrolled and/or clinically important pulmonary (including uncontrolled asthma), cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), hepatic, renal, endocrine (including Type 1 and Type 2 diabetes mellitus), hematologic, immunologic, neurologic, neurological (e.g., depression and/or anxiety disorders) or biliary disorders. Conditions which are well-controlled or resolved will be assessed by the Clinical Investigator on a case-by-case basis.
7. Uncontrolled hypertension determined by the blood pressure measured at Visit 1 (Day -7) and defined as (https://www.emedicinehealth.com/pediatric_vital_signs/article_em.htm):

   * Children 3-5 years old: Systolic blood pressure >107 mm Hg and diastolic blood pressure >71 mm Hg
   * Children 6-9 years old: Systolic blood pressure >110 mm Hg and diastolic blood pressure >73 mm Hg One re-test will be allowed on a separate day prior to Visit 2 (Day 0), for subjects whose blood pressure exceeds either of these cut points at Visit 1 (Day -7), in the judgment of the Clinical Investigator.
8. Extreme dietary habits as determined using the Diet Questionnaire (Appendix 2) and at the discretion of the Clinical Investigator.
9. History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
10. Major trauma or any other surgical event within 3 months of Visit 1 (Day -7).
11. Signs or symptoms of an active infection of clinical relevance within 5 days of Visit 1 (Day -7). The visit may be rescheduled such that all signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to Visit 1 (Day -7).*
12. Weight loss or gain >4.5 kg in the 3 months prior to Visit 1 (Day -7).
13. Currently or planning to be on a weight loss regimen during the study.
14. Antibiotic use within 3 months of Visit 1 (Day -7).
15. Use of steroids within 1 month of Visit 1 (Day -7).
16. Chronic use (i.e., daily on a regular basis) of anti-inflammatory medications (e.g., NSAIDs) within 1 month of Visit 1 (Day -7).
17. Use of medications (over-the-counter or prescription) and/or dietary supplements, known to influence GI function, including but not limited to prebiotics or probiotics, laxatives, enemas, fiber supplements and/or suppositories, antacids, anti-diarrheal agents, and/or anti-spasmodic within 2 weeks of Visit 1 (Day -7). Standard multivitamin and mineral supplements are allowed. Clinic staff will check ingredient lists of supplements for presence of prebiotics or probiotics.
18. Use of allergy medications (prescription or over the counter) for >2 times/week within 2 weeks of Visit 1 (Day -7).
19. Exposure to any non-registered drug product within 4 weeks prior to Visit 1 (Day -7).
20. Has a condition the Clinical Investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

    * If an infection occurs during the study period, test visits will be rescheduled until signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to study visits.

5.4.3 Excluded Products

* Antibiotics within 3 months of Visit 1 (Day -7) and throughout the study period.
* Steroids within 1 month of Visit 1 (Day -7) and throughout the study period.
* Chronic use (i.e., daily on a regular basis) of anti-inflammatory medications (e.g., NSAIDs) within 1 month of Visit 1 (Day -7) and throughout the study period.
* Medications (over-the-counter or prescription) and/or dietary supplements known to influence GI function, including but not limited to prebiotics or probiotics, laxatives, enemas, fiber supplements and/or suppositories, antacids, anti-diarrheal agents, and/or anti-spasmodic excluded within 2 weeks of Visit 1 (Day -7) and throughout the study period. Standard multivitamin and mineral supplements are allowed.
* Allergy medications of >2 times/week within 2 weeks of Visit 1 (Day -7). Consumption of any of these excluded products during the study period should be documented and subjects may be excluded from the Per Protocol population following a review of protocol deviations at the end of the intervention. Should a subject require any of these excluded products, the study staff should consult with the Clinical Investigator and/or designee to determine future action (e.g., early termination, extension of washout period, etc.)

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
GI Tolerance Composite Score | 10 day study period
  The electronic Bedtime GITQ contains a series of questions regarding the presence and severity of GI symptoms occurring from start of study product consumption in the morning until bedtime. The electronic Morning GITQ contains a series of questions regarding the presence and severity of GI symptoms occurring from bedtime until immediately prior to the consumption of study product the next morning. Individual GI symptoms include: gas/flatulence, abdominal cramping, abdominal distention/bloating, borborygmus/stomach rumbling, burping, and nausea and their severity is ranked on a 4-point scale ranging from none to severe.

SECONDARY OUTCOMES:
Effects of consuming soluble corn fiber on individual GI symptoms | Baseline, Days 1,2, 3,5,7 and 10 of each study product period.
  The electronic Bedtime GITQ contains a series of questions regarding the presence and severity of GI symptoms occurring from start of study product consumption in the morning until bedtime. The electronic Morning GITQ contains a series of questions regarding the presence and severity of GI symptoms occurring from bedtime until immediately prior to the consumption of study product the next morning. Individual GI symptoms include: gas/flatulence, abdominal cramping, abdominal distention/bloating, borborygmus/stomach rumbling, burping, and nausea and their severity is ranked on a 4-point scale ranging from none to severe.

OTHER OUTCOMES:
Dose response effects of soluble corn fiber on GI tolerance, stool consistency and bowel habits and fecal microbiome | up to 10 days
  Caregivers will be asked to help subjects complete an electronic BHD-BSS during the 3 days immediately prior to Visit 2 (Day 0) for collection of baseline information. Caregivers will also be asked to help subjects complete the BHD-BSS every day during the 10 days of study product consumption during each test period. If bowel movement occurs while the subject is not in close proximity to the caregiver (e.g., when subject is at school), the caregivers will be instructed to record the time of the bowel movement as best as possible, but not complete any other details (e.g., straining, consistency, etc) about that particular bowel movement. The diary will provide information on stool frequency and consistency, straining and discomfort during bowel movement, and any sensation of incomplete evacuation. Caregivers will be provided instructions on how to access the electronic BHD-BSS at Visit 1 (Day -7).
  Fecal samples will be collected using Omnigene®-GUT DNA Genotek per manufacturer's

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Kelley, Principal Investigator — Biofortis Innovation Services
Locations (1):
- Biofortis Innovation Services, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aziz I, Whitehead WE, Palsson OS, Tornblom H, Simren M. An approach to the diagnosis and management of Rome IV functional disorders of chronic constipation. Expert Rev Gastroenterol Hepatol. 2020 Jan;14(1):39-46. doi: 10.1080/17474124.2020.1708718. Epub 2020 Jan 2. PMID 31893959
- [Background] Boler BM, Serao MC, Bauer LL, Staeger MA, Boileau TW, Swanson KS, Fahey GC Jr. Digestive physiological outcomes related to polydextrose and soluble maize fibre consumption by healthy adult men. Br J Nutr. 2011 Dec;106(12):1864-71. doi: 10.1017/S0007114511002388. Epub 2011 May 31. PMID 21736814
- [Background] So D, Whelan K, Rossi M, Morrison M, Holtmann G, Kelly JT, Shanahan ER, Staudacher HM, Campbell KL. Dietary fiber intervention on gut microbiota composition in healthy adults: a systematic review and meta-analysis. Am J Clin Nutr. 2018 Jun 1;107(6):965-983. doi: 10.1093/ajcn/nqy041. PMID 29757343
- [Background] Ho J, Nicolucci AC, Virtanen H, Schick A, Meddings J, Reimer RA, Huang C. Effect of Prebiotic on Microbiota, Intestinal Permeability, and Glycemic Control in Children With Type 1 Diabetes. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4427-4440. doi: 10.1210/jc.2019-00481. PMID 31188437
- [Background] Housez B, Cazaubiel M, Vergara C, Bard JM, Adam A, Einerhand A, Samuel P. Evaluation of digestive tolerance of a soluble corn fibre. J Hum Nutr Diet. 2012 Oct;25(5):488-96. doi: 10.1111/j.1365-277X.2012.01252.x. Epub 2012 Jun 6. PMID 22672058
- [Background] Karalus M, Clark M, Greaves KA, Thomas W, Vickers Z, Kuyama M, Slavin J. Fermentable fibers do not affect satiety or food intake by women who do not practice restrained eating. J Acad Nutr Diet. 2012 Sep;112(9):1356-1362. doi: 10.1016/j.jand.2012.05.022. Epub 2012 Jul 6. PMID 22771185
- [Background] Klosterbuer AS, Hullar MA, Li F, Traylor E, Lampe JW, Thomas W, Slavin JL. Gastrointestinal effects of resistant starch, soluble maize fibre and pullulan in healthy adults. Br J Nutr. 2013 Sep 28;110(6):1068-74. doi: 10.1017/S0007114513000019. Epub 2013 Feb 7. PMID 23388502
- [Background] Klurfeld DM, Davis CD, Karp RW, Allen-Vercoe E, Chang EB, Chassaing B, Fahey GC Jr, Hamaker BR, Holscher HD, Lampe JW, Marette A, Martens E, O'Keefe SJ, Rose DJ, Saarela M, Schneeman BO, Slavin JL, Sonnenburg JL, Swanson KS, Wu GD, Lynch CJ. Considerations for best practices in studies of fiber or other dietary components and the intestinal microbiome. Am J Physiol Endocrinol Metab. 2018 Dec 1;315(6):E1087-E1097. doi: 10.1152/ajpendo.00058.2018. Epub 2018 Aug 21. PMID 30130151
- [Background] Molly K, Vande Woestyne M, Verstraete W. Development of a 5-step multi-chamber reactor as a simulation of the human intestinal microbial ecosystem. Appl Microbiol Biotechnol. 1993 May;39(2):254-8. doi: 10.1007/BF00228615. PMID 7763732
- [Background] Stewart ML, Nikhanj SD, Timm DA, Thomas W, Slavin JL. Evaluation of the effect of four fibers on laxation, gastrointestinal tolerance and serum markers in healthy humans. Ann Nutr Metab. 2010;56(2):91-8. doi: 10.1159/000275962. Epub 2010 Jan 19. PMID 20090313
- [Background] Timm DA, Thomas W, Boileau TW, Williamson-Hughes PS, Slavin JL. Polydextrose and soluble corn fiber increase five-day fecal wet weight in healthy men and women. J Nutr. 2013 Apr;143(4):473-8. doi: 10.3945/jn.112.170118. Epub 2013 Feb 20. PMID 23427334
- [Background] Van Hul M, Karnik K, Canene-Adams K, De Souza M, Van den Abbeele P, Marzorati M, Delzenne NM, Everard A, Cani PD. Comparison of the effects of soluble corn fiber and fructooligosaccharides on metabolism, inflammation, and gut microbiome of high-fat diet-fed mice. Am J Physiol Endocrinol Metab. 2020 Oct 1;319(4):E779-E791. doi: 10.1152/ajpendo.00108.2020. Epub 2020 Aug 24. PMID 32830554
- [Background] Whisner CM, Martin BR, Nakatsu CH, McCabe GP, McCabe LD, Peacock M, Weaver CM. Soluble maize fibre affects short-term calcium absorption in adolescent boys and girls: a randomised controlled trial using dual stable isotopic tracers. Br J Nutr. 2014 Aug 14;112(3):446-56. doi: 10.1017/S0007114514000981. Epub 2014 May 22. PMID 24848974
- See also: Institute of Medicine. Dietary Reference Intakes for Energy, Carbohydrates, Fiber, Fat, Fatty Acids, Cholesterol, Protein and Amino Acids. — https://www.nap.edu/read/10490/chapter/1
- See also: World Health Organization. Fact sheet: Diarrhoeal disease — https://www.who.int/en/news-room/fact-sheets/detail/diarrhoeal-disease